CLINICAL TRIAL: NCT04605094
Title: A Phase 2 Multinational, Randomized, Double-blind, Parallel-group, 16-week Placebo-controlled Study With a 36-Week Extension to Investigate the Use of Benralizumab for Patients With Moderate to Severe Atopic Dermatitis Despite Treatment With Topical Medications (The HILLIER Study)
Brief Title: Efficacy and Safety Study of the Use of Benralizumab for Patients With Moderate to Severe Atopic Dermatitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study did not meet the primary endpoint.
Sponsor: AstraZeneca (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D3256C00001
Record Dates: First submitted 2020-09-01; First posted 2020-10-27 (Actual); Results first posted 2023-06-27 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Atopic Dermatitis
Keywords: Moderate to severe atopic dermatitis; pruritus; skin lesion
MeSH Terms: conditions — Dermatitis, Atopic; Pruritus | interventions — benralizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Benralizumab (Experimental)
  Interventions: Biological: Benralizumab
- Placebo / Benralizumab (Experimental)
  Interventions: Biological: Placebo / Benralizumab

INTERVENTIONS:
Biological: Benralizumab — Benralizumab by subcutaneous injection until Week 16, and then benralizumab by subcutaneous injection during the extension period.
  Other Names: Benralizumab, Benra, Fasenra
  Arms: Benralizumab
Biological: Placebo / Benralizumab — Placebo by subcutaneous injection until Week 16, then benralizumab by subcutaneous injection until Week 52.
  Other Names: Benralizumab, Benra, Fasenra
  Arms: Placebo / Benralizumab

SUMMARY:
The purpose of the study is to compare the efficacy and safety of benralizumab versus placebo and to compare benralizumab dosing regimens during extension period.

DETAILED DESCRIPTION:
The aim of this study is to investigate the use of benralizumab as treatment for patients with moderate to severe atopic dermatitis (AD) who remain symptomatic despite treatment with topical medications. It is proposed that benralizumab will deplete eosinophils from affected skin, improve symptoms of AD, and improve AD-related quality of life. This Phase 2 study is designed to compare the efficacy of treatment with benralizumab versus placebo and compare benralizumab maintenance dosing regimens in the extension period.

ELIGIBILITY:
Inclusion Criteria:

1. Physician-confirmed diagnosis of AD (according to American Academy of Dermatology Consensus Criteria) that is not adequately controlled with topical medications.
2. EASI score of ≥ 12 at screening and ≥ 16 at randomization.
3. IGA score of ≥ 3 (on a scale of 0 to 4, in which 3 is moderate and 4 is severe) at screening and at randomization.
4. Atopic dermatitis involvement of ≥ 8% body- surface area at screening and ≥ 10% body-surface area at randomization.
5. A pruritus numerical rating scale average score for maximum itch intensity of ≥ 4, based on the average of daily pruritus numerical rating scale scores for maximum itch intensity reported during the 7 days prior to randomization.
6. Documented recent history (within 6 months prior to screening) of inadequate response to treatment with topical medications, or patients for whom topical treatments are otherwise medically inadvisable (eg, because of important side effects or safety risks).
7. Participants that have applied a stable dose of topical emollient (moisturizer) twice daily for ≥ 7 consecutive days immediately before the randomization visit. (NOTE: See exclusion criterion 11 for limitations regarding emollients)
8. Participants must be willing and able to complete daily PRO assessments:

   * Complete at least 70% of daily PRO assessments between Visit 1 and Visit 2 and
   * Complete at least 5 of 7 daily PRO assessments in the 7 days prior to Visit 2.
9. Females of childbearing potential (FOCBP) must agree to use a highly effective method of birth control (confirmed by the Investigator) from randomization, throughout the study duration, and within 16 weeks after last dose of IP and have a negative serum pregnancy test result on Visit 1.
10. Females not of childbearing potential are defined as females who are either permanently sterilized (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy) or who are postmenopausal. Females will be considered postmenopausal if they have been amenorrheic for ≥ 12 months prior to the planned date of randomization without an alternative medical cause. The following age-specific requirements apply:

    1. Females < 50 years old will be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatment and with follicle-stimulating hormone (FSH) levels in the postmenopausal range. Until FSH is documented to be within menopausal range, the participant should be treated as a FOCBP.
    2. Females ≥ 50 years old will be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatment.

Exclusion Criteria:

1. Participants with active dermatological conditions (eg, psoriasis, seborrheic dermatitis, cutaneous lymphoma) other than atopic dermatitis that, in the investigator's opinion, may interfere with the study assessments
2. Known active allergic or irritant contact dermatitis that, in the investigator's opinion, may interfere with the study assessments
3. Current malignancy, or history of malignancy, with the exception of:

   1. Participants who have had basal cell carcinoma, localized squamous cell carcinoma of the skin, or in situ carcinoma of the cervix are eligible provided that the participant is in remission and curative therapy was completed at least 12 months prior to the date informed consent, was obtained.
   2. Participants who have had other malignancies are eligible provided that the participant is in remission and curative therapy was completed at least 5 years prior to the date informed consent, was obtained.
4. Any disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, hematological, psychiatric, or major physical impairment that is not stable in the opinion of the Investigator and could:

   1. Affect the safety of the participant throughout the study
   2. Influence the findings of the studies or their interpretations
   3. Impede the participant's ability to complete the entire duration of study.
5. History of anaphylaxis to any biologic therapy or vaccine
6. A helminth parasitic infection diagnosed within 24 weeks prior to the date informed consent is obtained that has not been treated with, or has failed to respond to standard of care therapy
7. Any clinically significant abnormal findings in physical examination, vital signs, hematology, clinical chemistry, or urinalysis during screening/run-in period which, in the opinion of the Investigator, may put the participant at risk because of his/her participation in the study, or may influence the results of the study, or the participant's ability to complete entire duration of the study
8. Current active liver disease:

   1. Chronic stable hepatitis B and C (including positive testing for hepatitis B surface antigen [HBsAg] or hepatitis C antibody), or other stable chronic liver disease are acceptable if participant otherwise meets eligibility criteria. Stable chronic liver disease should generally be defined by the absence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice, or cirrhosis.
   2. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level ≥ 3 times the upper limit of normal (ULN), confirmed by repeated testing during the run-in period. Transient increase of AST/ALT level that resolves by the time of randomization is acceptable if in the Investigator's opinion the participant does not have an active liver disease and meets other eligibility criteria.
9. A history of known immunodeficiency disorder including a positive human immunodeficiency virus (HIV) test Prior/concomitant Therapy
10. Participants who have received treatment for AD with TCS, topical calcineurin inhibitors (TCI), or topical phosphodiesterase-4 (PDE4) inhibitors within the 7 days prior to the randomization visit
11. Initiation of treatment of AD with prescription moisturizers or moisturizers containing additives such as ceramide, hyaluronic acid, urea, or filaggrin degradation products during the screening period (patients may continue using stable doses of such moisturizers if initiated before the screening visit)
12. Regular use (2 visits per week) of a tanning booth/parlor or phototherapy for AD within 4 weeks prior to the randomization visit
13. Use of immunosuppressive medication including, but not limited to: methotrexate, cyclosporine, azathioprine, systemic corticosteroids within 4 weeks or 5 half-lives prior to the date informed consent is obtained, whichever is longer.

    Other
14. Receipt of immunoglobulin or blood products within 30 days prior to the date informed consent is obtained
15. Receipt of any marketed or investigational biologic within 4 months or 5 half-lives prior to the date informed consent is obtained, whichever is longer
16. Receipt of live attenuated vaccines 30 days prior to first dose of IP
17. Receipt of any investigational nonbiologic within 30 days or 5 half-lives prior to the date informed consent is obtained, whichever is longer
18. Previously received benralizumab (MEDI-563, FASENRA)
19. Change to allergen immunotherapy or new allergen immunotherapy within 30 days prior to the date of informed consent and anticipated changes in immunotherapy throughout the study
20. Planned elective major surgical procedures during the conduct of the study
21. Previous randomization in the present study
22. Concurrent enrollment in another clinical trial
23. AstraZeneca staff involved in the planning and/or conduct of the study
24. For females only: Currently pregnant, breastfeeding, or lactating females A serum pregnancy test will be done for FOCBP at Visit 1 and a urine pregnancy test must be performed for FOCBP at each subsequent treatment visit prior to IP administration. A positive urine test result must be confirmed with a serum pregnancy test. If serum test is positive, the participant should be excluded.

Ages: 12 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emma Guttman, MD, PhD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (42):
- United States (12):
  - Research Site, Los Angeles, California
  - Research Site, Newport Beach, California
  - Research Site, Bridgeport, Connecticut
  - Research Site, Fort Myers, Florida
  - Research Site, Tampa, Florida
  - Research Site, Ypsilanti, Michigan
  - Research Site, Portsmouth, New Hampshire
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Norman, Oklahoma
  - Research Site, Sugarloaf, Pennsylvania
- Australia (4):
  - Research Site, Kogarah
  - Research Site, Parkville
  - Research Site, Sippy Downs
  - Research Site, Woolloongabba
- Bulgaria (3):
  - Research Site, Haskovo
  - Research Site, Pleven
  - Research Site, Sofia
- Czechia (5):
  - Research Site, Brno
  - Research Site, Ostrava
  - Research Site, Ostrava-Poruba
  - Research Site, Pardubice
  - Research Site, Prague
- France (2):
  - Research Site, Brest
  - Research Site, Lille
- Poland (5):
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Osielsko
  - Research Site, Poznan
  - Research Site, Warsaw
- South Korea (6):
  - Research Site, Ansan-si
  - Research Site, Daegu
  - Research Site, Gwangju
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Yangsan
- Spain (5):
  - Research Site, Alicante
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Madrid
  - Research Site, Manises

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: HILLIER Brochure — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3256C00001&attachmentIdentifier=220141e8-ba2f-4aea-a044-80a5876025af&fileName=HILLIER_Brochure_V01_USA.pdf&versionIdentifier=
- See also: HILLIER Flyer — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3256C00001&attachmentIdentifier=b97b714c-8163-4691-b923-9d3cff3c16c6&fileName=HILLIER_Flyer_V01_USA.pdf&versionIdentifier=
- See also: HILLIER Patient Brochure — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3256C00001&attachmentIdentifier=5d60250f-ea3e-458b-8532-570d4c4a89c1&fileName=HILLIER_Patient_Brochure_V02_AUS(en)02.pdf&versionIdentifier=
- See also: HILLIER Patient Flyer — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3256C00001&attachmentIdentifier=8b961fc2-8fec-4c92-a573-9ea37c22a9cf&fileName=HILLIER_Patient_Flyer_V01_AUS(en).pdf&versionIdentifier=
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3256C00001&attachmentIdentifier=9411e493-5a39-4b9a-8a04-301ceccf1729&fileName=D3256C00001_Final_synopsis_CSR_Redacted_PDFA.pdf&versionIdentifier=
- See also: Statistical Analysis Plan (SAP) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3256C00001&attachmentIdentifier=b729f15f-82c5-448b-a10e-c0a9879bfc2c&fileName=D3256C00001_SAP_Final_Redacted_Final_PDFA.pdf&versionIdentifier=
- See also: Protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3256C00001&attachmentIdentifier=27a5a5f9-4d11-40b7-932c-2c742e598a11&fileName=D3256C00001-CSP_V3_Redacted_PDFA.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 2, double-blind, placebo-controlled study was conducted in participants with moderate to severe atopic dermatitis (AD) at 48 study centers in 8 countries.
Pre-assignment Details: This study consisted of a screening period (up to 4 weeks), placebo-controlled double-blind treatment period (up to 16 weeks) and an extension period (up to 36 weeks). A total of 194 participants were randomized and received treatment in this study.
Groups:
- Benralizumab: Participants received benralizumab 30 milligram (mg) subcutaneous (SC) injection on Day 1 visit for every 4 weeks (Q4W) until Week 16 visit. In extension phase, participants received benralizumab 30 mg SC injection for either Q4W or every 8 weeks (Q8W) until Week 52 visit.
- Placebo: Participants received placebo matching benralizumab on Day 1 visit for Q4W until Week 16. In extension phase, participants received benralizumab 30 mg SC injection for Q4W until Week 28 visit and then followed by benralizumab 30 mg SC injection for Q8W until Week 52 visit.
Period: Overall Study
Arm/Group | Benralizumab | Placebo
Started | 96 | 98
Completed | 37 | 37
Not Completed | 59 | 61
Not completed — Adverse Event | 2 | 2
Not completed — Lost to Follow-up | 1 | 4
Not completed — Physician Decision | 2 | 2
Not completed — Study terminated by Sponsor | 31 | 33
Not completed — Withdrawal by Subject | 22 | 19
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis set (FAS) consisted of all randomized participants who received at least 1 dose of study drug, irrespective of their protocol adherence and continued participation in the study.
Groups:
- Benralizumab: Participants received benralizumab 30 mg SC injection on Day 1 visit for Q4W until Week 16 visit. In extension phase, participants received benralizumab 30 mg SC injection for either Q4W or Q8W until Week 52 visit.
- Total: Total of all reporting groups
Arm/Group | Benralizumab | Placebo | Total
Number analyzed (Participants) | 96 | 98 | 194
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.8 (15.87) | 29.5 (16.00) | 29.6 (15.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 32 | 72
  Male | 56 | 66 | 122
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 6 | 6 | 12
  Asian | 24 | 20 | 44
  White | 65 | 70 | 135
  Other | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 13 | 24
  Not Hispanic or Latino | 85 | 85 | 170

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Investigator Global Assessment (IGA) 0/1 and a Decrease in IGA of ≥2 Points at Week 16 Relative to Baseline
Description: The IGA is an instrument used in clinical studies to rate the severity of AD globally, based on a 5-point scale ranging from 0 = clear; 1 = almost clear; 2 = mild disease; 3 = moderate disease; 4 = severe disease. The IGA used clinical characteristics of erythema, infiltration, papulation, oozing, and crusting as guidelines for the overall severity assessment. A higher score indicated greater severity. A responder at Week 16 was defined as having IGA 0/1 and a decrease in IGA of ≥2 points at Week 16 relative to baseline. Participants who withdrew from the study/required rescue therapy after Day 28 were considered as non-responders from the time these events occurred. Baseline was defined as the last recorded value on or prior to the date of randomization.
Time Frame: Baseline (Week 0) and at Week 16
Population: The FAS consisted of all randomized participants who received at least 1 dose of study drug, irrespective of their protocol adherence and continued participation in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 96 | 98
percentage of participants | 9.4 [3.36 to 14.93] | 17.3 [10.40 to 25.12]
Statistical Analysis 1: Comparison: Benralizumab vs Placebo; Treatment difference in IGA responders Estimates were from a logistic regression model that included treatment group, age as recorded on electronic case report form (eCRF) at screening (>=12 to <18 years; >=18 years), blood eosinophils as recorded on eCRF at screening (<300 cells/microliters [μL]; >=300 cells/μL) and baseline value of IGA score; Test type: Other; p = 0.080, Regression, Logistic; Difference in response rate = -8.62, 95% CI 2-sided [-17.94 to 0.71]

2. Secondary Outcome: Percentage of Participants Who Experienced 75% Reduction From Baseline in Eczema Area and Severity Index (EASI-75) at Week 16
Description: The EASI assessed the severity and extent of AD. Severity of 4 AD disease characteristics (erythema, induration/papulation, excoriation [scratching], lichenification) each were assessed on a scale of 0 (absent) to 3 (severe) in each of 4 body regions (head/neck, trunk, upper limbs, and lower limbs). Total body total score=sum of the region total scores; ranged from 0 to 72. Participants were classified as responders if they achieved at least 75% reduction from baseline in their EASI total score at Week 16. Participants who withdrew from study/required rescue therapy after Day 28 were non-responders from the time these events occurred. Higher scores indicated a more severe or more extensive condition. Baseline was defined as the last recorded value on or prior to the date of randomization.
Time Frame: Baseline (Week 0) and at Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 96 | 98
percentage of participants | 19.8 [11.71 to 27.45] | 24.5 [16.27 to 33.19]
Statistical Analysis 1: Comparison: Benralizumab vs Placebo; Treatment difference in EASI-75 responders Estimates were from a logistic regression model that included treatment group, age as recorded on eCRF at screening (>=12 to < 18 years; >=18 years), blood eosinophils as recorded on eCRF at screening (<300 cells/μL; >=300 cells/μL) and baseline EASI total score; Test type: Other; p = 0.384, Regression, Logistic; Difference in response rate = -5.15, 95% CI 2-sided [-16.67 to 6.36]

3. Secondary Outcome: Percentage of Participants Who Experienced 90% Reduction From Baseline in Eczema Area and Severity Index (EASI-90) at Week 16
Description: The EASI assessed the severity and extent of AD. Severity of 4 AD disease characteristics (erythema, induration/papulation, excoriation [scratching], lichenification) each were assessed on a scale of 0 (absent) to 3 (severe) in each of 4 body regions (head/neck, trunk, upper limbs, and lower limbs). Total body total score=sum of the region total scores; ranged from 0 to 72. Participants were classified as responders if they achieved at least 90% reduction from baseline in their EASI total score at Week 16. Participants who withdrew from study/required rescue therapy after Day 28 were non-responders from the time these events occurred. Higher scores indicated a more severe or more extensive condition. Baseline was defined as the last recorded value on or prior to the date of randomization.
Time Frame: Baseline (Week 0) and at Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 96 | 98
percentage of participants | 7.3 [2.05 to 12.42] | 15.3 [8.33 to 22.50]
Statistical Analysis 1: Comparison: Benralizumab vs Placebo; Treatment difference in EASI-90 responders Estimates were from a logistic regression model that included treatment group, age as recorded on eCRF at screening (>=12 to < 18 years; >=18 years), blood eosinophils as recorded on eCRF at screening (<300 cells/μL; >=300 cells/μL) and baseline EASI total score; Test type: Other; p = 0.078, Regression, Logistic; Difference in response rate = -8.18, 95% CI 2-sided [-16.94 to 0.59]

4. Secondary Outcome: Percentage of Participants With an Improvement of ≥4 or More Points in Peak Pruritus Weekly Score
Description: The peak pruritus numeric rating scale (NRS) was a 1-item daily assessment of the worst itch the participant experienced over the past 24 hours. The score ranged from 0 to 10, with 0 being "no itch" and 10 being "worst itch imaginable" and so a reduction in score was considered an improvement. A responder was defined as having an improvement of 4 or more points relative to baseline. Participants who withdrew from the study/required rescue therapy after Day 28 were considered as non-responders from the time these events occurred. The Week 16 weekly scores were defined as the average of the daily scores for the 7 days prior to the weekly score.
Time Frame: At Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 96 | 98
percentage of participants | 14.6 [7.87 to 21.70] | 14.3 [7.28 to 20.90]
Statistical Analysis 1: Comparison: Benralizumab vs Placebo; Treatment difference in Peak Pruritus NRS Estimates were from a logistic regression model that included treatment group, age as recorded on eCRF at screening (>=12 to < 18 years; >=18 years), blood eosinophils as recorded on eCRF at screening (<300 cells/μL; >=300 cells/μL) and baseline Peak Pruritus score; Test type: Other; p = 0.889, Regression, Logistic; Difference in response rate = 0.69, 95% CI 2-sided [-8.93 to 10.32]

ADVERSE EVENTS:
Time Frame: Adverse events in the on-study period were reported from the first dose of study treatment (Day 1) up to end of follow-up, approximately a maximum up to Week 60
Description: The Safety Analysis set consisted of all participants who received at least 1 dose of study drug.
Groups:
- Placebo: Participants received placebo matching benralizumab on Day 1 visit for Q4W until Week 16 in placebo-controlled treatment period.
- Placebo to Benralizumab: Participants who completed placebo-controlled treatment period entered extension phase. Participants received benralizumab 30 mg SC injection for Q4W until Week 28 visit and then followed by benralizumab 30 mg SC injection for Q8W until Week 52 visit.
Arm/Group | Benralizumab | Placebo | Placebo to Benralizumab
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/98 | 0/87
Serious Adverse Events (participants affected / at risk) | 3/96 | 0/98 | 2/87
Other Adverse Events (participants affected / at risk) | 38/96 | 10/98 | 29/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benralizumab (N=96) | Placebo (N=98) | Placebo to Benralizumab (N=87)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paranasal sinus inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benralizumab (N=96) | Placebo (N=98) | Placebo to Benralizumab (N=87)
Bronchitis (Infections and infestations) | 5 (5) | 0 (0) | 4 (4)
Conjunctivitis (Infections and infestations) | 3 (4) | 0 (0) | 6 (6)
COVID-19 (Infections and infestations) | 21 (23) | 4 (4) | 14 (14)
Nasopharyngitis (Infections and infestations) | 9 (10) | 0 (0) | 7 (8)
Upper respiratory tract infection (Infections and infestations) | 9 (12) | 2 (3) | 5 (5)
Headache (Nervous system disorders) | 4 (4) | 5 (8) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated as the study did not support the continued development of benralizumab for the indication of AD.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/94/NCT04605094/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-16): https://cdn.clinicaltrials.gov/large-docs/94/NCT04605094/SAP_001.pdf